CLINICAL TRIAL: NCT05976399
Title: The Investigation of The Effectiveness Of Manual Lymph Drainage in Individuals With Migraine
Brief Title: Manual Lymph Drainage in Individuals With Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Özlem Çınar Özdemir, Assoc. prof, Izmir Democracy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MLD in Migraine
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Manual Lymphatic Drainage
Keywords: Migraine; Manual Lymphatic Drainage; Connective Tissue Massage; Quality of Life
MeSH Terms: conditions — Migraine Disorders | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Intervention Model Description: The study included forty individuals with migraine. Participants' neck pain was evaluated with the Neck Pain and Disability Scale, pressure perceptions and pain sensitivity with an algometer, quality of life with the Short Form-3, and headaches with a pain diary kept for 15 days before and after treatment. Then, the individuals were randomly divided into two as the manual lymph drainage group and the connective tissue massage group. Both groups were treated for 45 minutes twice a week for 6 weeks. The groups were assessed before the treatment and at the end of 6 weeks.
Who Masked: Participant
Masking Description: The individuals to be included in the study were listed on the computer according to their application order, and then a randomization process was employed to divide them into two groups: the manual lymph drainage group and the connective tissue massage group. Individuals with odd-numbered positions were assigned to the manual lymph drainage group, while individuals with even-numbered positions were assigned to the connective tissue massage group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual lymph drainage group (Active Comparator): The patients, who had filled out their pain diary before and submitted a consent form, were first evaluated before the treatment and then they lay on their back with their neck area open, paying attention to the protection of their privacy. Hand strokes, one of the basic techniques applied for treatment, were planned in accordance with the anatomy and physiology of the lymphatic system. MLD was applied to the lateral neck and face region in 5-7 repetitions so that the lymph collectors could give an adequate reaction to the application. The treatment was performed 2 days a week for 6 weeks, with a total of 12 sessions. Each session lasted 45 minutes.
  Interventions: Other: Manual Lymph Drainage
- Connective tissue massage group (Active Comparator): In participants in the CTM group, the treatment was started with the sacral region called the "basic region" and the whole back was treated. Pulls in the interscapular region were more intense than in other regions. After the interscapular region, the cervical, clavicular, and facial regions were also included in the treatment. The applications first started with the basic region and then progressed to the lower thoracic, scapular, and interscapular regions. Then, the cervical and clavicular regions were treated. In each region, the applications were performed three times on each of the right and left sides. While positioning the patients, we paid attention to their privacy and the temperature of the room where the treatment was carried out. A total of 12 sessions, which were conducted 2 days a week and took 6 weeks, were performed.
  Interventions: Other: Connective Tissue Massage

INTERVENTIONS:
Other: Connective Tissue Massage — In participants in the CTM group, the treatment was started with the sacral region called the "basic region" and the whole back was treated. Pulls in the interscapular region were more intense than in other regions. After the interscapular region, the cervical, clavicular, and facial regions were also included in the treatment. Both short and long pulls were used according to the region during CTM. The applications first started with the basic region and then progressed to the lower thoracic, scapular, and interscapular regions. Then, the cervical and clavicular regions were treated. In each region, the applications were performed three times on each of the right and left sides. While positioning the patients, we paid attention to their privacy and the temperature of the room where the treatment was carried out. A total of 12 sessions, which were conducted 2 days a week and took 6 weeks, were performed.
  Arms: Connective tissue massage group
Other: Manual Lymph Drainage — The patients, who had filled out their pain diary before and submitted a consent form, were first evaluated before the treatment and then they lay on their back with their neck area open, paying attention to the protection of their privacy. Hand strokes, one of the basic techniques applied for treatment, were planned in accordance with the anatomy and physiology of the lymphatic system. MLD was applied to the lateral neck and face region in 5-7 repetitions so that the lymph collectors could give an adequate reaction to the application. The treatment was performed 2 days a week for 6 weeks, with a total of 12 sessions. Each session lasted 45 minutes.
  Arms: Manual lymph drainage group

SUMMARY:
In the literature, research into the examination of the effect of MLD on migraine is quite limited. Our study aimed to examine the effectiveness of manual lymph drainage and connective tissue massage treatments on neck pain and disability, sleep quality, pain threshold and severity, depression and quality of life.

DETAILED DESCRIPTION:
Although there are evidence-based guidelines for clinical decision-making and reporting the care of patients with migraine, migraine management for the population is inadequate. Even among individuals who are correctly diagnosed, almost more than half of patients are not administered any acute or preventive treatment. Various invasive and non-invasive treatment options are available in the treatment of migraine. Relaxation training, exercise, cold application, massage, transcutaneous electrical nerve stimulation (TENS), biofeedback, manipulation and mobilization techniques, and trigger point therapy are some of the non-invasive treatment options used in migraine treatment. These treatments, which can be applied independently, can also be applied in combination with pharmacological treatments in some patients. In addition, the patient's knowledge about the disease makes it easier to manage the process and cope with the pain better.

Connective tissue massage (CTM) is a manipulative therapy method that is different from traditional massages in terms of both technical and physiological effects and has been used for diagnosis or treatment since 1928. Although the manipulative procedures applied target superficial connective and subcutaneous tissues, they also have effects on organs far from the local stimulation area. Another approach to migraine prophylaxis includes manual lymph drainage (MLD). It is considered that MLD causes sympathetic and parasympathetic effects and is similar to therapeutically effective relaxation therapy by reducing the hyperexcitability of the central system. With the parasympathetic effect it creates, it helps to reduce muscle pain and spasm, making it easier to cope with tension and stress. Reduction of the tension and stress factors may reduce the triggering of migraine and make it easier to cope with the current migraine. Recent studies have shown that the meningeal lymphatic system is located in the brain and that this system is a new way for the drainage of the cerebrospinal fluid.

In the literature, research into the examination of the effect of MLD on migraine is quite limited. We planned this randomized controlled trial to contribute to the reduction of pain and increase the quality of life of individuals with migraine by increasing the awareness of individuals working in this field in our country.

ELIGIBILITY:
Inclusion Criteria:

* To be able to read and write
* Diagnosis of migraine by a neurologist according to IHS criteria
* Be willing to participate in the study voluntarily signing an informed consent form
* Have good cognitive functioning
* Between the ages of 18 and 65
* Reported pain intensity of 40 mm or more according to VAS
* Headache (without allodynia) <15 days per month

Exclusion Criteria

* Had any of the contraindications of MLD for the general and neck region
* Had a history of neuromuscular disease,
* Had communication problems to the extent that prevented evaluation methods,
* Had headaches lasting >15 days a month, were diagnosed with other types of headaches (cervicogenic type headache, tension-type headache),
* Were diagnosed with fibromyalgia or myofascial pain syndrome, exhibited whiplash and similar traumas
* Had severe depression symptoms according to the Beck depression inventory,
* Had a congenital musculoskeletal anomaly, received non-pharmacological migraine treatment (acupuncture, dry needling, etc.),

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Pressure algometer (Dolorimeter) | All individuals participating in the study were evaluated before and after the 6-week-long treatment
  The pressure algometer was developed by Fischer to determine the perception of pressure and assess pain sensitivity. in our study, measurements with a dolorimeter were made from a total of 12 regions, including 6 on the right and 6 on the left. Selected 6 muscles were M. Temporalis anterior, M. Sternocleidomastoid, M. Scalenous anterior, M. Suboccipital, M. Levator scapula, and M. Trapezius (Upper).

SECONDARY OUTCOMES:
Neck Pain and Disability Scale | All individuals participating in the study were evaluated before and after the 6-week-long treatment
  It consists of 20 questions that examine the relationship between the severity of neck pain and social, functional, and emotional status. The questions on the scale are scored between 0 and 5 points. A high score indicates severe disability in patients.
Visual Analog Scale | All individuals participating in the study were evaluated before and after the 6-week-long treatment
  The severity of individuals' pain was evaluated using the visual analog scale. The patient evaluates his or her subjective pain sensation with this scale. It is a 100-mm-long horizontal or vertical scale, where 0 indicates no pain and 10 indicates the most severe pain possible
Pain diary | in the study a pain diary were given 2 weeks before the initiation of treatment and after the 6-week-long treatment was completed
  This is a method that is used to plan treatment and determine its effectiveness. It includes a diary in which the patient records information, such as the onset of pain, its severity, location, factors that increase or decrease it, and the name and dose of the medication used if any. Forty patients with migraine who were planned to be included in the study were given a pain diary 2 weeks before the initiation of treatment. Patients were asked to record the severity and duration of the pain, the symptoms accompanying it, and the name and the number of medications taken in the pain diary when they had a headache.
Short Form-36 | All individuals participating in the study were evaluated before and after the 6-week-long treatment
  This form was developed by Ware Jr and Sherbourne to evaluate the quality of life.It consists of 36 items that measure 8 dimensions: physical functioning, role limitations due to physical problems, social functioning, role limitations due to emotional problems, pain, mental health, the general perception of health, and energy/vitality. The dimensions are independent of each other, and a high score indicates the quality of life for that dimension.
Back Depression Inventory | All individuals participating in the study were evaluated before and after the 6-week-long treatment
  he Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression.
The Pittsburgh Sleep Quality Index | All individuals participating in the study were evaluated before and after the 6-week-long treatment
  The Pittsburgh Sleep Quality Index is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Çinar Özdemir, Assoc.Dr, Study Director — Izmir Democracy University; Betül Yıldırım, Principal Investigator — Siirt University
Locations (1):
- Izmir Democracy University, Izmir, Karabağlar/İZMİR, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goadsby PJ, Holland PR, Martins-Oliveira M, Hoffmann J, Schankin C, Akerman S. Pathophysiology of Migraine: A Disorder of Sensory Processing. Physiol Rev. 2017 Apr;97(2):553-622. doi: 10.1152/physrev.00034.2015. PMID 28179394
- [Background] Goats GC, Keir KA. Connective tissue massage. Br J Sports Med. 1991 Sep;25(3):131-3. doi: 10.1136/bjsm.25.3.131. PMID 1777777
- [Background] Happe S, Peikert A, Siegert R, Evers S. Erratum to: The efficacy of lymphatic drainage and traditional massage in the prophylaxis of migraine: a randomized, controlled parallel group study. Neurol Sci. 2016 Oct;37(10):1753. doi: 10.1007/s10072-016-2657-z. No abstract available. PMID 27412032
- [Derived] Yildirim Bulut B, Cinar Ozdemir O. Comparison of the efficacy of connective tissue massage and manual lymphatic drainage in patients with migraine: a randomized controlled trial. J Oral Facial Pain Headache. 2025 Sep;39(3):121-132. doi: 10.22514/jofph.2025.054. Epub 2025 Sep 12. PMID 41070573